CLINICAL TRIAL: NCT01295788
Title: Simultaneous vs Delayed Initiation of REAL-Time Continuous Glucose Monitoring in Children and Adolescents With Type 1 Diabetes Starting Insulin Pump Therapy
Brief Title: Timing of Initiation of Continuous Glucose Monitoring in Established Pediatric Diabetes (The CGM TIME Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Canadian Clinical Trial Network (Unknown)
Responsible Party: Principal Investigator, Margaret Lawson, Professor of Pediatrics, Children's Hospital of Eastern Ontario
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHEO 09/05E
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Simultaneous or Delayed initiation of continuous glucose monitoring
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simultaneous RT-CGM and Pump Initiation (Experimental): The experimental group will initiate RT-CGM at the same time as they begin insulin pump therapy.
  Interventions: Device: Simultaneous RT-CGM and Pump Initiation
- Delayed RT-CGM Initiation (Active Comparator): The control group will use standard pump therapy until the 6 month study visit at which time RT-CGM will be initiated.
  Interventions: Device: Delayed Initiation of RT-CGM

INTERVENTIONS:
Device: Simultaneous RT-CGM and Pump Initiation — Subjects in this group will start using RT-CGM at the same time as they initiate insulin pump therapy.
  Other Names: Sensor-Augmented Pump Therapy at Pump Initiation
  Arms: Simultaneous RT-CGM and Pump Initiation
Device: Delayed Initiation of RT-CGM — Subjects in this group will start using RT-CGM 6 months after initiation of insulin pump therapy.
  Arms: Delayed RT-CGM Initiation

SUMMARY:
The investigators hypothesize that REAL-Time Continuous Glucose Monitoring (RT-CGM) will be more effective if introduced in children and adolescents with established diabetes at the same time as they are starting pump therapy. This randomized controlled trial will compare the effectiveness of simultaneous vs delayed introduction of RT-CGM in children and adolescents with type 1 diabetes who are starting insulin pump therapy.

DETAILED DESCRIPTION:
REAL-Time Continuous Glucose Monitoring (RT-CGM) improves diabetes control in adults with type 1 diabetes. However, studies of RT-CGM in children and adolescents have been mostly negative. The lack of effectiveness in the pediatric population appears directly related to adherence to RT-CGM, i.e., the willingness of children and teens to wear and use this technology. Most previous RT-CGM studies have focused on experienced pump users or children with new-onset diabetes. At the time of pump initiation, children and adolescents who have been living with diabetes (and their parents) are highly motivated to make changes in their diabetes management and to take on additional responsibilities to improve their diabetes control and lifestyle, the two primary reasons for initiating pump therapy in the pediatric population. The investigators hypothesize that readiness for making changes in diabetes management will be greater at the time of pump initiation than at six months after the pump start. Further, the investigators hypothesize that readiness for change at the time of RT-CGM initiation will predict future adherence to RT-CGM and its effectiveness.

ELIGIBILITY:
Inclusion criteria:

* Males and females age 5-18 years old.
* Established T1D diagnosis for a minimum of one year.
* Naïve to CSII therapy and ready to start CSII with the Veo pump (Medtronic) .
* Willing to use RT-CGM and to be randomly assigned to either simultaneous or delayed RT-CGM initiation.
* Regular diabetes follow up at one of the 5 participating sites.
* Internet access at home (to upload RT-CGM data).
* Parent(s) or legally acceptable representative able to speak and read English or French.
* Ability of the subject and parent(s) or legally acceptable representative to participate in all aspects of this clinical trial.
* Written informed consent must be obtained and documented, with assent of the child if <14 years of age.

Exclusion Criteria

* Conditions which in the opinion of the investigator may interfere with the subject's ability to participate in the study.
* Has received oral and/or intravenous steroid therapy (for any indication, at any dose and/or for any duration) on more than 2 separate occasions in the past 12 months. Use of inhaled and/or topical steroid therapy in the last 12 months does not exclude the subject.
* Prior use of RT-CGM for more than 50% of the time over the past 6 months.
* Prior enrollment in the current study.
* Current enrollment in another intervention trial.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Adherence to CGM (hours per week) | one year
  Number of hours of RT-CGM use per week

SECONDARY OUTCOMES:
A1C | one year
  Hemoglobin A1C
Readiness for change | six months
  SOCRATES - Diabetes Version
Treatment Satisfaction and Quality of Life | one year
  Insulin Delivery Systems Rating Questionnaire (IDSRQ)
Fear of Hypoglycemia | one year
  Hypoglycemia Fear Scale (HFS-98)
Barriers to Adherence | one year
  Modified Barriers to Adherence Questionnaire (MBAQ)
Perception of Barriers/Facilitators to RT-CGM Use | one year
  CGM Satisfaction Scale (CGM-SAT)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L Lawson, MD, Study Director — Children's Hospital of Eastern Ontario
Locations (5):
- Canada (5):
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Markham-Stouffville Hospital, Markham, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lawson ML, Verbeeten KC, Courtney JM, Bradley BJ, McAssey K, Clarson C, Kirsch S, Curtis JR, Mahmud FH, Richardson C, Cooper T, Chan J, Tang K. Timing of CGM initiation in pediatric diabetes: The CGM TIME Trial. Pediatr Diabetes. 2021 Mar;22(2):279-287. doi: 10.1111/pedi.13144. Epub 2020 Nov 4. PMID 33098212
- [Result] Verbeeten KC, Perez Trejo ME, Tang K, Chan J, Courtney JM, Bradley BJ, McAssey K, Clarson C, Kirsch S, Curtis JR, Mahmud FH, Richardson C, Cooper T, Lawson ML; CGM TIME Trial Study Group and the JDRF Canadian Clinical Trials Group. Fear of hypoglycemia in children with type 1 diabetes and their parents: Effect of pump therapy and continuous glucose monitoring with option of low glucose suspend in the CGM TIME trial. Pediatr Diabetes. 2021 Mar;22(2):288-293. doi: 10.1111/pedi.13150. Epub 2020 Nov 27. PMID 33179818
- [Derived] Lawson ML, Bradley B, McAssey K, Clarson C, Kirsch SE, Mahmud FH, Curtis JR, Richardson C, Courtney J, Cooper T, Downie CJ, Rajamannar G, Barrowman N; CGM TIME Trial Study Group; JDRF Canadian Clinical Trial Network CCTN1101. The JDRF CCTN CGM TIME Trial: Timing of Initiation of continuous glucose Monitoring in Established pediatric type 1 diabetes: study protocol, recruitment and baseline characteristics. BMC Pediatr. 2014 Jul 18;14:183. doi: 10.1186/1471-2431-14-183. PMID 25034216
- [Derived] Olivier P, Lawson ML, Huot C, Richardson C, Nakhla M, Romain J. Lessons learned from a pilot RCT of simultaneous versus delayed initiation of continuous glucose monitoring in children and adolescents with type 1 diabetes starting insulin pump therapy. J Diabetes Sci Technol. 2014 May;8(3):523-8. doi: 10.1177/1932296814524855. Epub 2014 Feb 27. PMID 24876616